CLINICAL TRIAL: NCT04166890
Title: Comparison of the Efficacy and Safety of Two Homologous Active Principles for Local Dental Anesthesia: Non-inferiority Trial
Brief Title: Comparison of the Efficacy and Safety of Two Homologous Active Principles for Local Dental Anesthesia
Acronym: ECA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Principal Investigator, Germán David Arboleda Toro, Assistant Professor, Universidad de Antioquia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: Ensayo Clinico Articaina
Record Dates: First submitted 2019-10-08; First posted 2019-11-18 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Drug Effect; Tooth Extraction
Keywords: Articaine; IANB; Third molar surgery; Non-inferiority; Local anesthesia
MeSH Terms: interventions — Carticaine

STUDY DESIGN:
Intervention Model Description: Open, randomized, double blind, controlled, phase 4 crossover, randomized clinical trial will be conducted to compare the efficacy and clinical safety of two homologous active principles, articaine HCl with 1: 100,000 epinephrine (test) against the reference formulation 4% articaine HCl with 1: 100,000 of epinephrine, used intraorally in extraction of retained third molars (18), and will be carried out in the Faculty of Dentistry of the University of Antioquia
Who Masked: Participant, Care Provider, Investigator
Masking Description: Both anesthetics will be masked so that no differences are observed between them at the time of their application by the surgeon, clinical monitor and patient. Therefore, they will be covered with adhesive paper marked with the letter A or B. Each pair of anesthetics will be stored in an envelope and inside it will say the side that would apply each anesthetic (right or left) and each envelope will have a consecutive number from 1 to 196, and will be delivered to each patient in order of arrival at the study.
  Being a double blind study, it must be guaranteed that neither the patient, nor the surgeon, nor the clinical monitor knows about the allocation of treatments at the time of intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- NS Lower right molar (Experimental): IANB Artheek SP Articaine EPINEPHrine Cartridge 4% 1:100000
  Interventions: Drug: Articaine / EPINEPHrine Cartridge
- SD Lower Left molar (Active Comparator): IANB Septanest Articaine EPINEPHrine Cartridge 4% 1:100000
  Interventions: Drug: Articaine / EPINEPHrine Cartridge
- NS Lower left molar (Experimental): IANB Artheek SP Articaine EPINEPHrine Cartridge 4% 1:100000
  Interventions: Drug: Articaine / EPINEPHrine Cartridge
- SD Lower right molar (Active Comparator): IANB Septanest Articaine EPINEPHrine Cartridge 4% 1:100000
  Interventions: Drug: Articaine / EPINEPHrine Cartridge

INTERVENTIONS:
Drug: Articaine / EPINEPHrine Cartridge — The day scheduled for the surgery, vital signs (pulse, blood pressure and oxygen saturation) will be recorded prior the administration of the anesthesia. A volume of 1.8 ml of 4% articaine and epinephrine 1: 100000 solution of either the test product or the reference product will be deposited slowly to proceed to the inferior alveolar nerve block (IANB), according to the table of allocation of treatments in each period. The vital signs will continue to be monitored during the procedure, and once the procedure has been completed. If the volunteer needs more anesthetic, this will be recorded and will be administrated according to the maximum permitted doses (7 mg / kg (up to 500 mg) 5 mg / kg in children 7), and immediately after the administration, the vital signs will be taken again.

SUMMARY:
In the complexity of the Dental care the third molar surgery is one of the most common procedures, it is indicated for multiple reasons like infections in root canal, prosthetics or even esthetical purposes. This surgery can be safely performed with the help of local anesthetics, due to their quick action, and reversibility to control pain, reducing possible complications during and after the surgeries.

Among the different types of local anesthetics used in dentistry, the articaine bears characteristics that provide some advantages compared to similar anesthetics like Lidocaine, being one of the most used anesthetics worldwide. Different authors have concluded that it is a safe when used in patients at different ages and it is effective as a local anesthetic in the majority of procedures. It is important for dentists to know the differences or similarities of anesthetics in terms of their effects, safety, dosages required in patients undergoing surgical removal of teeth, as well as the mechanism of action and pharmacological properties, in order to take advantage of its benefits and minimize risks.

This study aims to test the efficacy and safety of an anesthetic solution, based on the same active molecule, articaine, manufactured by two different commercial houses, one domestic and one international, in order to gather scientific evidence and to show that they are not different. This will provide scientific results to help in the selection of any of these brands to be used with confidence in the dental practice. This will strengthen the collaboration between the academy and the companies, which would allow them to improve the quality of their products.

Locally there are no studies available comparing the articaine-type anesthetic with epinephrine at the same concentration, manufactured locally by a national company, to a foreign one, which is an important opportunity to expand the knowledge and create scientific reports, about what a local anesthetic is and what it does.

Finally, this study would contribute to the need to guarantee the quality of medicines in Colombia, by means of compliance with the legal provisions contemplated in resolution 1890 of November 2001 and 1400 of August 2001, issued by the Ministry of Health of Colombia : "Requirements to demonstrate the therapeutic effectiveness, through studies of Bioavailability and Bioequivalence of medicines for a special group of them.

DETAILED DESCRIPTION:
Local anesthetic:

Local anesthetics are widely used in dentistry for different procedures and are chemical substances that block nerve conduction, temporarily and irreversibly in order to avoid pain and are placed in specific sites of the body, for example in oral tissues.

Pharmacology of local anesthetics related to effectiveness and safety

Latency time It is defined as the time that elapses between the infiltration of the anesthetic substance in the tissue until the first signs of insensibility are felt. It is influenced by the distance of the route the anesthetic must travel, with the ability to cross the membrane of the nerve cells.

Duration of the anesthetic effect Also known as the duration of the action, related to the capacity of fixation of the anesthetic substance to the nerve cell proteins and with lipid solubility.

pH of anesthetics It is one of the factors that influence the action of blocking nerve conduction, and is the factor that conditions the movement of the anesthetic from the site where it is administered to the nerve fiber, that is why the tissues that are infected make the effectiveness is decreased, since the pH would turn acidic. In addition, the pH varies according to whether or not it has a vasoconstrictor.

Power Anesthetic capacity to pass the lipids of the nerve membranes, the greater the liposolubility, the greater the anesthetic power, depending on how the power is the classification of the action time, low power with short action, intermediate power with action medium and high power with long action.

Diffusion It is related to the minimum concentration required to inhibit nerve conduction, given by the transfer of molecules or ions from an anesthetic solution from the point where it infiltrates to the membrane of the nerve cell.

Articaine

Articaine is a short-acting local anesthetic, belonging to the group of amides, it has an additional ester group that is rapidly hydrolyzed by plasma esterases, which exhibits a lower toxicity compared to other drugs of the same family. This dissolves better than other amides in the soft tissues and bone, for this reason, it is especially indicated for dental use.

Articaine is introduced in 1972 in the market of local anesthetics. Prepared for the first time by Rusching et al in 1969, it changed its generic name to articaine when it began to be used in clinical practice in Germany in 1976. Its use gradually expanded, until it entered the market of the United States and Canada, in 1983 and in the United Kingdom in 1998.

Articaine with vasoconstrictor (epinephrine) is administered submucosally. The onset of anesthetic effects is observed between 1 to 6 minutes and the duration of anesthesia is approximately one hour and is recommended for long procedures. After administration, maximum concentrations are reached after 20 minutes, approximately between 60 and 80% bind plasma proteins, in particular albumin and gamma globulins, and are easily distributed in soft tissues.

Its main metabolite is the articainic acid, which is metabolized by the isoenzymes of the cytochrome P450, between 5 and 10% of the articainic acid; this causes the increase of the elimination, half-life to 90 minutes. The drug is eliminated in the urine as articainic acid, as glucuronide of the articainic acid and as articaine without metabolizing.

The administration of vasoconstrictors such as epinephrine, together with an anesthetic, could cause increases in blood pressure or heart rate due to higher plasma levels, however, these adverse effects are uncommon.

Patients receiving local anesthesia for dental treatments may experience side effects at the level of the Central Nervous System (CNS), in case of receiving an intra-arterial injection with reflux into the cerebral circulation. Patients with peripheral vascular diseases and hypertension may experience an exaggerated response when treated with articaine-epinephrine due to the vasoconstrictive effects of epinephrine, which can be especially intense in the elderly.

Because of its bisulfite content (as a preservative of epinephrine), the preparations of articaine-epinephrine are contraindicated in patients with hypersensitivity to bisulfite. In addition, patients with asthma are usually more susceptible than others to this hypersensitivity.

There are few studies evaluating the pharmacokinetics of articaine in the elderly or in patients with renal or hepatic insufficiency, although caution is advised when administering articaine-epinephrine to patients with liver diseases, as these patients are more susceptible to the drug's potential toxicity and Dose reductions may be necessary. It should also be administered with caution in patients with a history of drug abuse because the adverse reactions are dose-related and in elderly patients should be dosed with the minimum effective dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women, criteria assessed during anamnesis
* Age between 18 and 25 years old
* Presence of lower third molars in the mouth with no level of eruption determined by the clinical oral examination
* Weight / height ratio with a coefficient of variation of no more than 15% of the ideal weight, according to the tables of the Metropolitan Life Insurance
* Lower third molars in a mesio-angulated position evidenced by the panoramic radiography taken for the study in the Faculty of Dentistry of the University of Antioquia, and which is in Nolla's stage equal or greater than 6
* Voluntary acceptance to participate in the study by signing the informed consent

Exclusion Criteria:

* Presence of phobias or traumas related to the dental practice and/or with needles
* Presence of clinical problems such as kidney diseases, cardiovascular diseases, known allergies or drug hypersensitivity discovered through the anamnesis of the clinical history prepared for the investigation
* Hi consumption of alcohol or cigarettes
* Presence of problems related to drug dependence
* Being ill for the last two weeks before the study begins
* use of enzyme inhibitors or inducers for four weeks prior to the participation in the study
* Have used any medication or natural product, seven days prior to the first part of the study
* Have donated blood in the last three months
* Have participated in another clinical trial, thirty days prior to the first part of the study
* Be a member of the research group or a relative of the responsible personnel involved in the study.

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 179 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Number of patients with total absence of sensitivity and pain | 2 to 8 minutes
  Assessment of total absence of tactile and pain sensitivity after administration of the anesthetics.
Failure | 10 minutes
  Assessment of the inability to block tactile sensitivity or painful sensitivity
Pain assessed by visual analogue pain scale | One hour (1h)
  Monitoring of the visual analogue pain (VAS) scale, where the amount of pain patient feels ranges from 0, non pain to 10, extreme amount of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Fabian Jaimes, MD, PhD, Study Director — Universidad de Antioquia
Locations (1):
- University of Antioquia, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim C, Hwang KG, Park CJ. Local anesthesia for mandibular third molar extraction. J Dent Anesth Pain Med. 2018 Oct;18(5):287-294. doi: 10.17245/jdapm.2018.18.5.287. Epub 2018 Oct 31. PMID 30402548
- [Background] Castañeda DA, Briceño CR, Sánchez AE, Rodrí- guez A, Castro D, Barrientos S. Prevalencia de dientes incluidos, retenidos e impactados analizados en radiografías panorámicas de población de Bogotá, Colombia. Univ Odontol. 2015 Jul-Dic; 34(73): 149-157. http://dx.doi.org/10.11144/ Javeriana.uo34-73.
- [Background] Organización Mundial de la Salud (OMS). Marco Conceptual de la Clasificación Internacional para la Seguridad del Paciente. Ginebra: OMS; 2009.
- [Background] Becker DE, Reed KL. Essentials of local anesthetic pharmacology. Anesth Prog. 2006 Fall;53(3):98-108; quiz 109-10. doi: 10.2344/0003-3006(2006)53[98:EOLAP]2.0.CO;2. PMID 17175824
- [Background] Aggarwal V, Singla M, Miglani S, Kohli S. Efficacy of Articaine Versus Lidocaine Administered as Supplementary Intraligamentary Injection after a Failed Inferior Alveolar Nerve Block: A Randomized Double-blind Study. J Endod. 2019 Jan;45(1):1-5. doi: 10.1016/j.joen.2018.09.012. Epub 2018 Dec 6. PMID 30527595
- [Background] St George G, Morgan A, Meechan J, Moles DR, Needleman I, Ng YL, Petrie A. Injectable local anaesthetic agents for dental anaesthesia. Cochrane Database Syst Rev. 2018 Jul 10;7(7):CD006487. doi: 10.1002/14651858.CD006487.pub2. PMID 29990391
- [Background] Mittal J, Kaur G, Mann HS, Narang S, Kamra M, Kapoor S, Sindhi M, Kataria R. Comparative Study of the Efficacy of 4% Articaine vs 2% Lidocaine in Surgical Removal of Bilaterally Impacted Mandibular Third Molars. J Contemp Dent Pract. 2018 Jun 1;19(6):743-748. PMID 29959306
- [Result] Snoeck M. Articaine: a review of its use for local and regional anesthesia. Local Reg Anesth. 2012;5:23-33. doi: 10.2147/LRA.S16682. Epub 2012 Jun 5. PMID 22915899
- [Result] Bartlett G, Mansoor J. Articaine buccal infiltration vs lidocaine inferior dental block - a review of the literature. Br Dent J. 2016 Feb 12;220(3):117-20. doi: 10.1038/sj.bdj.2016.93. PMID 26868800
- [Result] Meechan JG. How to overcome failed local anaesthesia. Br Dent J. 1999 Jan 9;186(1):15-20. doi: 10.1038/sj.bdj.4800006. PMID 10028738
- [Result] Vree TB, Gielen MJ. Clinical pharmacology and the use of articaine for local and regional anaesthesia. Best Pract Res Clin Anaesthesiol. 2005 Jun;19(2):293-308. doi: 10.1016/j.bpa.2004.12.006. PMID 15966499
- [Result] Katyal V. The efficacy and safety of articaine versus lignocaine in dental treatments: a meta-analysis. J Dent. 2010 Apr;38(4):307-17. doi: 10.1016/j.jdent.2009.12.003. Epub 2009 Dec 16. PMID 20006669
- [Result] Malamed SF, Gagnon S, Leblanc D. Efficacy of articaine: a new amide local anesthetic. J Am Dent Assoc. 2000 May;131(5):635-42. doi: 10.14219/jada.archive.2000.0237. PMID 10832257
- [Result] Suresh K. An overview of randomization techniques: An unbiased assessment of outcome in clinical research. J Hum Reprod Sci. 2011 Jan;4(1):8-11. doi: 10.4103/0974-1208.82352. PMID 21772732
- [Result] Hersh EV, Giannakopoulos H, Levin LM, Secreto S, Moore PA, Peterson C, Hutcheson M, Bouhajib M, Mosenkis A, Townsend RR. The pharmacokinetics and cardiovascular effects of high-dose articaine with 1:100,000 and 1:200,000 epinephrine. J Am Dent Assoc. 2006 Nov;137(11):1562-71. doi: 10.14219/jada.archive.2006.0092. PMID 17082283
- [Result] Haas DA. An update on local anesthetics in dentistry. J Can Dent Assoc. 2002 Oct;68(9):546-51. PMID 12366885
- [Result] Haase A, Reader A, Nusstein J, Beck M, Drum M. Comparing anesthetic efficacy of articaine versus lidocaine as a supplemental buccal infiltration of the mandibular first molar after an inferior alveolar nerve block. J Am Dent Assoc. 2008 Sep;139(9):1228-35. doi: 10.14219/jada.archive.2008.0338. PMID 18762633
- [Derived] Arboleda-Toro D, Toro L, Osorio-Osorno YA, Castrillon-Pino L, Florez-Zapata NMV. Comparing Articaine brands: A randomized non-inferiority controlled trial. Heliyon. 2021 Jun 9;7(6):e07252. doi: 10.1016/j.heliyon.2021.e07252. eCollection 2021 Jun. PMID 34195402